CLINICAL TRIAL: NCT01142349
Title: Cognitive Behavioral Therapy for Arthritis Pain and Insomnia in Older Adults
Acronym: Lifestyles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Michael Vitiello, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01AG031126 (NIH); R01AG031126 (NIH)
Record Dates: First submitted 2010-05-26; First posted 2010-06-11 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Pain Dysfunction; Sleep Disturbance; Osteoarthritis
Keywords: Arthritis; Group Program; Pain; Insomnia; Pain dysfunction and sleep disturbance among older adults with osteoarthritis.
MeSH Terms: conditions — Parasomnias; Osteoarthritis; Arthritis; Pain; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lifestyles A (Experimental): Cognitive Behavioral Therapy for Pain and Insomnia
  Interventions: Behavioral: Lifestyles A
- Lifestyle B (Experimental): Cognitive Behavioral Therapy for Pain
  Interventions: Behavioral: Lifestyles B
- Lifestyles C (Active Comparator): Osteoarthritis Education
  Interventions: Behavioral: Lifestyles C

INTERVENTIONS:
Behavioral: Lifestyles A — Six weekly group sessions that last about 90-120 minutes presenting cognitive behavioral therapy for pain and insomnia
  Arms: Lifestyles A
Behavioral: Lifestyles B — Six weekly group sessions that last about 90-120 minutes presenting cognitive behavioral therapy for pain.
  Arms: Lifestyle B
Behavioral: Lifestyles C — Six weekly group sessions that last about 90-120 minutes presenting osteoarthritis education.
  Arms: Lifestyles C

SUMMARY:
This study compares the efficacy of three group interventions for people with co-morbid osteoarthritis (OA) and insomnia to help them manage their OA symptoms. The investigators hypothesize that a combination cognitive-behavioral treatment will produce significantly greater initial and long-term improvements in OA symptoms than will the other two treatments.

DETAILED DESCRIPTION:
This study is only for members of the Group Health Cooperative (GHC) of Puget Sound who have both osteoarthritis pain and insomnia. The first part of the study involves filling out a mailed survey. Based on the results of the survey some respondents will be eligible for the second part of the study. Our goal in the second part is to test three different treatments for managing OA symptoms. The programs teach about things people with arthritis can do to improve the quality of their lives. All three programs deal with pain, sleep, mood and activity-but each has a slightly different focus. Participants will be randomly assigned to one of the three programs. Each program is made up of six weekly group sessions that last about 90-120 minutes. The programs will be co-led by licensed therapists and each will include 8-12 members. Study participants will also take part in a series of visits at their homes over the next 18 months. At each visit the investigators will ask them to do a few other study activities, such as keep a 7-day diary of their sleep and fill out a survey about their arthritis pain. With their permission the investigators will also ask them to let us collect some information from their GHC medical records.

ELIGIBILITY:
Inclusion Criteria:

* Age 60+
* Continuously enrolled in Group Health one year prior to sample pull
* Primary care clinic at selected clinics
* Not in "No Contact File"
* Diagnosis 715xx (Osteoarthritis) in prior three years

Exclusion Criteria:

* Not continuously enrolled in Group Health for at least one year
* Medical record information indicates a diagnosis of:

  1. rheumatoid arthritis
  2. obstructive sleep apnea
  3. periodic leg movement disorder
  4. restless leg syndrome
  5. sleep-wake cycle disturbance
  6. rapid eye movement (REM) behavior disorder
  7. dementia or receiving cholinesterase inhibitors
  8. Parkinson's disease or other neurodegenerative disease known to directly impact sleep
  9. cancer in the past year and receiving chemotherapy or radiation therapy in the past year
  10. inpatient treatment for congestive heart failure within the previous 6 months

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 367 (Actual)
Dates: Start 2009-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | Baseline
  A 7-item self-report screening measure that rates severity of sleep problems, interference with daily functioning, and participant distress over symptoms. Rated on a scale from 0 (no problems) to 4 (very much a problem).
Insomnia Severity Index (ISI) | Post treatment- 2 months post baseline assessment
  A 7-item self-report screening measure that rates severity of sleep problems, interference with daily functioning, and participant distress over symptoms. Rated on a scale from 0 (no problems) to 4 (very much a problem).
Insomnia Severity Index (ISI) | 9 months post baseline assessment
  A 7-item self-report screening measure that rates severity of sleep problems, interference with daily functioning, and participant distress over symptoms. Rated on a scale from 0 (no problems) to 4 (very much a problem).
Insomnia Severity Index (ISI) | 18 months post baseline assessment
  A 7-item self-report screening measure that rates severity of sleep problems, interference with daily functioning, and participant distress over symptoms. Rated on a scale from 0 (no problems) to 4 (very much a problem).
Global Pain Severity-Graded Chronic Pain Scale | Baseline
  The Global Pain Severity Scale derived from the Graded Chronic Pain Scale consists of three 0-10 pain intensity ratings (pain right now, average pain, and worst pain in the prior month) and three 0-10 pain interference ratings (interference with daily activities, recreational, social and family activites, and ability to work including housework).
Global Pain Severity-Graded Chronic Pain Scale | Post treatment-2 mos. post baseline
  The Global Pain Severity Scale derived from the Graded Chronic Pain Scale consists of three 0-10 pain intensity ratings (pain right now, average pain, and worst pain in the prior month) and three 0-10 pain interference ratings (interference with daily activities, recreational, social and family activites, and ability to work including housework).
Global Pain Severity-Graded Chronic Pain Scale | 9 months post baseline assessment
  The Global Pain Severity Scale derived from the Graded Chronic Pain Scale consists of three 0-10 pain intensity ratings (pain right now, average pain, and worst pain in the prior month) and three 0-10 pain interference ratings (interference with daily activities, recreational, social and family activites, and ability to work including housework).
Global Pain Severity- Graded Chronic Pain Scale | 18 months post baseline assessment
  The Global Pain Severity Scale derived from the Graded Chronic Pain Scale consists of three 0-10 pain intensity ratings (pain right now, average pain, and worst pain in the prior month) and three 0-10 pain interference ratings (interference with daily activities, recreational, social and family activites, and ability to work including housework).

CONTACTS AND LOCATIONS:
Overall Officials: Michael V Vitiello, Ph.D., Principal Investigator — University of Washington; Susan M McCurry, Ph.D., Principal Investigator — University of Washington; Michael Von Korff, Sc.D., Principal Investigator — Group Health Research Institute; Ben Balderson, Ph.D., Principal Investigator — Group Health Research Institute
Locations (2):
- United States (2):
  - Group Health Research Institute, Seattle, Washington
  - University of Washington, Seattle, Washington

REFERENCES:
- [Background] Smith MT, Haythornthwaite JA. How do sleep disturbance and chronic pain inter-relate? Insights from the longitudinal and cognitive-behavioral clinical trials literature. Sleep Med Rev. 2004 Apr;8(2):119-32. doi: 10.1016/S1087-0792(03)00044-3. PMID 15033151
- [Background] Smith MT, Edwards RR, McCann UD, Haythornthwaite JA. The effects of sleep deprivation on pain inhibition and spontaneous pain in women. Sleep. 2007 Apr;30(4):494-505. doi: 10.1093/sleep/30.4.494. PMID 17520794
- [Background] Moffitt PF, Kalucy EC, Kalucy RS, Baum FE, Cooke RD. Sleep difficulties, pain and other correlates. J Intern Med. 1991 Sep;230(3):245-9. doi: 10.1111/j.1365-2796.1991.tb00438.x. PMID 1895046
- [Background] Rybarczyk B, Stepanski E, Fogg L, Lopez M, Barry P, Davis A. A placebo-controlled test of cognitive-behavioral therapy for comorbid insomnia in older adults. J Consult Clin Psychol. 2005 Dec;73(6):1164-74. doi: 10.1037/0022-006X.73.6.1164. PMID 16392989
- [Background] Montgomery P, Dennis J. Cognitive behavioural interventions for sleep problems in adults aged 60+. Cochrane Database Syst Rev. 2002;2003(2):CD003161. doi: 10.1002/14651858.CD003161. PMID 12076472
- [Derived] Thakral M, Von Korff M, McCurry SM, Morin CM, Vitiello MV. ISI-3: evaluation of a brief screening tool for insomnia. Sleep Med. 2021 Jun;82:104-109. doi: 10.1016/j.sleep.2020.08.027. Epub 2020 Aug 27. PMID 33910159
- [Derived] Vitiello MV, McCurry SM, Shortreed SM, Baker LD, Rybarczyk BD, Keefe FJ, Von Korff M. Short-term improvement in insomnia symptoms predicts long-term improvements in sleep, pain, and fatigue in older adults with comorbid osteoarthritis and insomnia. Pain. 2014 Aug;155(8):1547-1554. doi: 10.1016/j.pain.2014.04.032. Epub 2014 May 1. PMID 24793909
- [Derived] McCurry SM, Shortreed SM, Von Korff M, Balderson BH, Baker LD, Rybarczyk BD, Vitiello MV. Who benefits from CBT for insomnia in primary care? Important patient selection and trial design lessons from longitudinal results of the Lifestyles trial. Sleep. 2014 Feb 1;37(2):299-308. doi: 10.5665/sleep.3402. PMID 24497658
- [Derived] Vitiello MV, McCurry SM, Shortreed SM, Balderson BH, Baker LD, Keefe FJ, Rybarczyk BD, Von Korff M. Cognitive-behavioral treatment for comorbid insomnia and osteoarthritis pain in primary care: the lifestyles randomized controlled trial. J Am Geriatr Soc. 2013 Jun;61(6):947-956. doi: 10.1111/jgs.12275. Epub 2013 May 27. PMID 23711168